CLINICAL TRIAL: NCT02000011
Title: Interest of a Geriatric Intervention Plan Associated to a Comprehensive Geriatric Assessment on Autonomy, Quality of Life and Survival of Patients Aged 70 Years Old and More Surgically Treated for a Resectable Cancer (Thoracic, Digestive or Urologic). Randomized Multicentric Study
Acronym: epigac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-A01038-37; 2013-33 (Other: AP HM)
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Cancer
Keywords: patients; aged 70 years old; thoracic,; digestive or; urological; resectable
MeSH Terms: conditions — Neoplasms | interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard strategy (Other)
  Interventions: Other: comprehensive geriatric assessment (CGA)
- experimental strategy (Experimental)
  Interventions: Other: comprehensive geriatric assessment (CGA); Other: Geriatric intervention plan (GIP)

INTERVENTIONS:
Other: comprehensive geriatric assessment (CGA)
Other: Geriatric intervention plan (GIP)
  Arms: experimental strategy

SUMMARY:
The curative treatment of thoracic (lung and oesophagus), digestive (gastric, pancreatic, hepatic, colorectal), and urologic (renal, bladder, prostatic) cancers needs a surgical resection. For patients aged of 70 years old and more, this surgery is associated to an increased morbid-mortality especially because of more frequent co-morbidities. Comprehensive geriatric assessment (CGA) allows distinguishing patients for whom a resection surgery can be complicated by high morbid-mortality or a loss of autonomy. It has been proved that for old patient population without cancer, CGA associated with a geriatric intervention plan (GIP) allows autonomy preservation, decrease of institution admission, and survival improvement. The reference study showed that a CGA associated to a GIP improves survival of old patients who had a cancer surgery. However this study included patients from 60 years old and the GIP consisted in 3 home visits and 5 phone calls during the 4 weeks following hospital discharge.

We propose to perform a prospective and randomized study to evaluate the impact of a CGA with GIP in 70 years old and more patients with a thoracic, digestive or urologic cancer resection, respectively 1, 3, 6 and 12 months after discharge. CGA and GIP will focus on 8 distinct fields: autonomy, co-morbidities, co-medication, mobility, nutritional status, depression, cognitive function and social status. The impact of such a strategy on autonomy and survival has never been studied.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 70 years old or more
* Patient with a resectable cancer( thoracic, digestive ore urologic);
* Patients who have to undergo a surgery with general anaesthesia;
* Patients treated in one of the partner programme unit ;
* Patient able to fill in an auto-questionnaire alone or with some help;
* Patient who have signed an informed consent and who commits himself or herself to respect the protocol instructions.

Exclusion Criteria:

* Patient younger than 70 years old;
* Patient who is not registered to the social ;
* Patient for whom surgery is performed under local anaesthesia;
* Patient unable to fill-in alone an autoquestionnaire (because of an inability to read French language or severe cognitive troubles);
* Patient treated with neuroleptic or lithium ;
* Patient with already known cognitive impairment (Alzheimer, dementia, neurologic sequel);
* Patient under legal protection;
* Patient who has not signed informed consent.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2016-04-18 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
the 6-month autonomy after surgery | 24 MONTHS

SECONDARY OUTCOMES:
12-month autonomy | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France